CLINICAL TRIAL: NCT02968290
Title: Quantification of Posterior Capsule Opacity With Software Analysis Comparing Intraocular Lenses Hydrophilic x Hydrophobic in Pediatric Cataracts
Brief Title: Quantification of Posterior Capsule Opacification in Pediatric Cataract
Acronym: Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, camila ribeiro koch pena, Professor of medical residency of ophthalmology and PhD student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: University od São Paulo
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Posterior Capsule Opacification
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrofobic material-Alcon AcrySof SA60AT (Active Comparator): Intervention- Cataract Surgery with implantation of intraocular lens. In this arm will be implantation hydrofobic material.
  Interventions: Procedure: Cataract Surgery; Device: Alcon AcrySof SA60AT
- Hydrophilic material-Bausch Lomb AkreosA (Active Comparator): Intervention- Cataract Surgery with implantation of intraocular lens. In this arm will be implantation hydrophilic material.
  Interventions: Procedure: Cataract Surgery; Device: Bausch Lomb AkreosA

INTERVENTIONS:
Procedure: Cataract Surgery — Implant of intraocular lens hydrophobic or Implant of intraocular lens hydrophilic (Device)
Device: Alcon AcrySof SA60AT — Implant of intraocular lens hydrophobic
  Arms: Hydrofobic material-Alcon AcrySof SA60AT
Device: Bausch Lomb AkreosA — Implant of intraocular lens hydrophilic
  Arms: Hydrophilic material-Bausch Lomb AkreosA

SUMMARY:
The purpose of this study is to quantify the opacity of posterior capsule in pediatric cataract comparing two intraocular lens materials.

DETAILED DESCRIPTION:
The eye exam at the first appointment will consist of anamnesis, external motor, evaluating strabismus and nystagmus, visual acuity with and without correction, biomicroscopy, fundoscopy, binocular ultrasound biometry, pachymetry and specular microscopy. The surgery will be performed by a single surgeon under general anesthesia. All participants will receive primary intraocular lens implantation as the randomization process, or hydrophobic acrylic material or hydrophilic acrylic. The implanted intraocular lens differ primarily in the material. The lens of hydrophobic acrylic materials (AcrySof SA60AT, Alcon Lab) single, folding part, material acrylate / methacrylate with UV protection AcrySof filter, optical diameter of 6.0 mm, total length of 13.0 mm, haptic angle of 0 degree with 360 degree double square edge, spherical convex earlier. The lens hydrophilic acrylic material (Akreos ADAPT, Bausch and Lomb) single, folding piece with optical diameter 6.00 mm and length de10.7 mm aspheric convex in anterior and posterior with absorbent UV, haptic angle 0 degree angulation . It has 4 attachment points (haptics) with 360 degree square double edge.

ELIGIBILITY:
Inclusion Criteria:

* indication for cataract surgery

Exclusion Criteria:

* traumatic cataract
* neurological diseases that do not allow the exams

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Opacification of posterior capsule measured by graduation through the software EPCO software | 360 days after cataract surgery
  Photodocumentation with camera coupled to slit lamp adapter with external coaxial illumination of a fiber optic cable to the camera. After, analysis of opacification of the posterior capsule through the Evaluation of Posterior Capsule opacification software (EPCO 2000). The EPCO (Evaluation of Posterior Capsule Opacification) software is commercially available and offers some free access. The individual PCO score is calculated by multiplying the density of the opacification by the fraction of capsule area involved behind the IOL optic. It graded the PCO as 0 (none), 1 (minimal), 2 (mild), 3 (moderate) or 4 (severe). EPCO is one of the most used software for this purpose.

CONTACTS AND LOCATIONS:
Locations (1):
- Humberto Castro Lima, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Resnikoff S, Pascolini D, Etya'ale D, Kocur I, Pararajasegaram R, Pokharel GP, Mariotti SP. Global data on visual impairment in the year 2002. Bull World Health Organ. 2004 Nov;82(11):844-51. Epub 2004 Dec 14. PMID 15640920
- [Result] Gasper C, Trivedi RH, Wilson ME. Complications of Pediatric Cataract Surgery. Dev Ophthalmol. 2016;57:69-84. doi: 10.1159/000442502. Epub 2016 Apr 1. PMID 27043393
- [Result] Panahi-Bazaz MR, Zamani M, Abazar B. Hydrophilic Acrylic versus PMMA Intraocular Lens Implantation in Pediatric Cataract Surgery. J Ophthalmic Vis Res. 2009 Oct;4(4):201-7. PMID 23198075
- [Result] Lin H, Yang Y, Chen J, Zhong X, Liu Z, Lin Z, Chen W, Luo L, Qu B, Zhang X, Zheng D, Zhan J, Wu H, Wang Z, Geng Y, Xiang W, Chen W, Liu Y; CCPMOH Study Group. Congenital cataract: prevalence and surgery age at Zhongshan Ophthalmic Center (ZOC). PLoS One. 2014 Jul 3;9(7):e101781. doi: 10.1371/journal.pone.0101781. eCollection 2014. PMID 24992190
- [Result] Werner L, Tetz M, Feldmann I, Bucker M. Evaluating and defining the sharpness of intraocular lenses: microedge structure of commercially available square-edged hydrophilic intraocular lenses. J Cataract Refract Surg. 2009 Mar;35(3):556-66. doi: 10.1016/j.jcrs.2008.11.042. PMID 19251151
- [Result] Kleinmann G, Zaugg B, Apple DJ, Bleik J. Pediatric cataract surgery with hydrophilic acrylic intraocular lens. J AAPOS. 2013 Aug;17(4):367-70. doi: 10.1016/j.jaapos.2013.04.007. Epub 2013 Aug 6. PMID 23928003